CLINICAL TRIAL: NCT02541253
Title: An Open-label(Part1), Single Arm(Part1), Randomized(Part2), Double-blind(Part2), Active-controlled(Part2), Phase III Study to Evaluate the Efficacy and Safety of 'GC3110A(QIV)' in Healthy Children
Brief Title: A Study to Evaluate the Efficacy and Safety of 'GC3110A(QIV)' in Healthy Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GC3110A_C_P3
Record Dates: First submitted 2015-08-28; First posted 2015-09-04 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GC3110A (Experimental): One injection : 0.5ml or 0.25ml, IM on day 0 Two injection : 0.5ml or 0.25ml, IM on day 0
  Interventions: Biological: GC3110A
- GCFLU Pre-filled Syringe inj. (Active Comparator): One injection : 0.5ml or 0.25ml, IM on day 0 Two injection : 0.5ml or 0.25ml, IM on day 0
  Interventions: Biological: GCFLU Pre-filled Syringe inj.

INTERVENTIONS:
Biological: GC3110A — A single 0.5mL dose intramuscular injection
  Arms: GC3110A
Biological: GCFLU Pre-filled Syringe inj. — A single 0.5mL dose intramuscular injection
  Arms: GCFLU Pre-filled Syringe inj.

SUMMARY:
1. Part 1 If study subject and legal guardians who decide voluntarily to participate the clinical trial, and sign the Informed Consent Form (In the case of study subject less than 7 years of age, written informed consent by study subject's legal guardians), study subjects eligible for participating this trial protocol were assigned to test group and receiving the test drug 1 times or 2 times according to age.
2. Part 2 If study subject and legal guardians who decide voluntarily to participate the clinical trial, and sign the Informed Consent Form(In the case of study subject less than 7 years of age, written informed consent by study subject's legal guardians), the study subjects eligible for participating this trial protocol were assigned to test group or control group with the ratio of 4:1 and receiving the test drug 1 times or 2 times according to age as below;

   * 6 m ~ 3 years
   * 3 years ~ 9 years
   * 9 years ~ 19 years

DETAILED DESCRIPTION:
1. Part 1 If study subject and legal guardians who decide voluntarily to participate the clinical trial, and sign the Informed Consent Form (In the case of study subject less than 7 years of age, written informed consent by study subject's legal guardians), study subjects eligible for participating this trial protocol were assigned to test group and receiving the test drug 1 times or 2 times according to age.

   The safety data collected during part A will be reviewed by DSMB to evaluate the solicited adverse events for 7 days after each vaccination.

   However, if no toxicity higher than grade 3 according to FDA guidance the study was allowed to proceed to Part 2 without DSMB review.

   Efficacy and safety assessment methods, and visiting schedule will be the same as Part 2.
2. Part 2 If study subject and legal guardians who decide voluntarily to participate the clinical trial, and sign the Informed Consent Form(In the case of study subject less than 7 years of age, written informed consent by study subject's legal guardians), the study subjects eligible for participating this trial protocol were assigned to test group or control group with the ratio of 4:1 and receiving the test drug 1 times or 2 times according to age as below;

   * 6 m ~ 3 years
   * 3 years ~ 9 years
   * 9 years ~ 19 years The investigator will evaluate the efficacy and safety of the test product while clinical trial.

Blood samples will be collected at visit 1 for efficacy evaluation. The study subject and their legal guardians will be educated to daily record AEs after vaccination on the patient diary to evaluate the safety.

At visit1, blood samples will be collected from randomized study subjects and investigational drug of doses of 0.25mL or 0.5mL according to age will be intramuscularly injected. However, those who had not been vaccinated with influenza vaccine, aged of over than 6 months to less than 9 years study subjects, will re-visit and have the 2nd vaccination, 4~5 weeks after the 1st vaccination.

After 4~5 weeks since last vaccination, study subjects will visit and blood sample will be collected. And the serious adverse events occurred during 180 days after the final vaccination will be checked through the telephone visit.

The study subjects with 1 dose of vaccine will have 4 visits including Visit 1~2 and Visit 5~6. The study subjects with 2 dose of vaccine will have 6 visits including Visit 1~2, Visit 3~4 and Visit 5~6.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants and adolescents aged 6 month to 19 years
2. study Subject was born at full term pregnancy(37 weeks)
3. study Subject who understand the details of this clinical trial, decide voluntarily to participate the trial, and signed the Informed Consent Form (less than 7 years of age, written informed consent by study subject's legal guardians)

Exclusion Criteria:

1. Those with a history of allergic reaction to eggs or chicken, the vaccine components
2. Those who had been ad ministered the influenza vaccine 6 months prior to the study drug vaccination
3. Those with immunologic impairment including immune deficiency disorders or family history about it.
4. Those with a history of Guillain-Barre syndrome
5. Those with a history of Down's syndrome or cytogenetic disorders
6. Those who would be ineligible to participate the study as follows: serious chronic disease (cardiovascular system disease; excluding controlled hypertension and respiratory system disease; including respiratory failure, metabolic disease, renal dysfunction, hemoglobinopathy, etc)
7. Hemophilia patients at risk of serious bleeding with intramuscular injection or those receiving anticoagulant therapy
8. Those who have active infection or who have fever higher than 38.0℃ within 72 hours prior to the dosing of study drug
9. Those who had been vaccinated with another vaccine within 28 days prior to the dosing of study drug or had a scheduled vaccination during the clinical trial period
10. Those who had received an immunosuppressant, immunity-modifying drug within 3 months prior to the dosing of study drug - (1) Azathioprine, Cyclosporin, Interferon, G-CSF, Tacrolimus, Everolimus, Sirolimus, etc., (2) Those receiving high dose of corticosteroid(15mg/day of prednisolone is acceptable, but study subject used consistently 2mg/kg more than 14days is considered a high dose, so excluded in this clinical trial. However, inhalated, intra nasal and topical administration is acceptable regardless of dose.
11. Those who had received immunoglobulin or a blood-derived product within 3 months prior to the dosing of study drug or is scheduled to receive those products during the study period
12. Those who had taken antipyretic/analgesic/nonsteroidal antiinflammatory drugs within 4 hours prior to the dosing of study drug
13. study Subject who had participated in other clinical trial within 28 days prior to the study vaccination
14. Those whose clinically significant medical or psychiatric condition at the discretion of the investigator that would be ineligible to participate the study

Ages: 6 Months to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 543 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The percentage of study subjects achieving seroconversion* for HI antibody(seroconversion rate) The percentage of study subjects achieving a post-vaccination HI antibody titer≥1:40 (seroprotection rate) | Post-vaccination (Day 28)
  the percentage of study subjects with a pre-vaccination (Day 0) HI titer<1:10 and post-vaccination (Day 28) HI antibody titer≥1:40(Case1), or the percentage of study subjects with a pre-vaccination HI antibody titer≥1:10 and a minimum four-fold rise in post-vaccination HI antibody titer(Case 2)

SECONDARY OUTCOMES:
GMT | Post-vaccination (Day 28)
  GMT (Geometric Mean Titer) of HI antibody titer before vaccination (Day 0) and after vaccination (Day 28)
GMR | Post-vaccination (Day 28)
  GMR (Geometric Mean Ratio) of HI antibody titer before vaccination (Day 0) and after vaccination (Day 28)
The solicited adverse events (7 days after vaccination) | Post-vaccination (Day 7)
  The presence of the solicited adverse events occurred during 7 days after vaccination Local reaction: pain, tenderness, erythema/redness, induration/swelling Systemic reaction: fever, sweating, chills, nausea/vomiting, diarrhea, fatigue/malaise, headache, myalgia, arthralgia
The unsolicited adverse events (28 days after vaccination) | Post-vaccination (Day 28)
  The presence of the unsolicited adverse events occurred during 28 days after the study vaccination

OTHER OUTCOMES:
SAEs (VIsit 1 to Day 180) | VIsit 1 (Day 0) to Day 180
  The presence of the serious adverse events occurred from visit 1 to day 180

CONTACTS AND LOCATIONS:
Overall Officials: Jin-han Kang, Dr., Principal Investigator — The Catholic Univ. of Korea Seoul St. Mary's Hospital
Locations (12):
- South Korea (12):
  - Changwon Fatima Hospital, Changwon
  - Keimyung University Dongsan Medical Center, Daegu
  - The Catholic Univ. of Korea Daejeon St. Mary's Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Eulji University Medical Center, Seoul
  - Kepco Medical Center, Seoul
  - Korea Cancer Center Hospital, Seoul
  - The Catholic Univ. of Korea Seoul St. Mary's Hospital, Seoul
  - The Catholic Univ. of Korea St. Vincent's Hospital, Suwon
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee J, Lee KY, Kim JH, Kim CS, Eun BW, Kim HM, Kim DH, Hong YJ, Choi YY, Jo DS, Ma SH, Kang JH. Safety and Immunogenicity of an Egg-Cultivated Quadrivalent Inactivated Split-virion Influenza Vaccine (GC3110A) in Healthy Korean Children: a Randomized, Double-blinded, Active-controlled Phase III Study. J Korean Med Sci. 2018 Mar 26;33(13):e100. doi: 10.3346/jkms.2018.33.e100. PMID 29573247